CLINICAL TRIAL: NCT04525404
Title: MOIST Study: Multi-Organ Imaging With Serial Testing in COVID-19 Infected Patients
Acronym: MOIST
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Collaborators: Canadian VIGOUR Centre (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00102389
Record Dates: First submitted 2020-08-17; First posted 2020-08-25 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2022-09

CONDITIONS: Covid19; Coronavirus Infection; SARS-CoV Infection
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Severe Acute Respiratory Syndrome | interventions — Magnetic Resonance Imaging; Neuropsychological Tests; Spirometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Troponin Substudy: Participants with new COVID-19 infection will undergo high-sensitivity Troponin testing; participants with elevated Troponin will undergo MRI, bloodwork, and olfaction testing at Baseline, then repeat MRI, bloodwork and all functional testing at the Recovered (ie 12weeks post diagnosis) phase. Participants with normal Troponin will undergo only olfaction testing and bloodwork at baseline, then MRI, bloodwork and all functional testing at the Recovered phase.
  Interventions: Diagnostic Test: MRI (heart, brain, lungs, liver); Diagnostic Test: Bloodwork; Other: Cognitive testing; Other: Olfaction testing; Diagnostic Test: Spirometry; Other: Walk Test
- Late Cross-Sectional Substudy: Participants with a COVID-19 diagnosis at least 3 months prior to enrollment will undergo MRI, bloodwork and all functional testing at the Recovered phase only.
  Interventions: Diagnostic Test: MRI (heart, brain, lungs, liver); Diagnostic Test: Bloodwork; Other: Cognitive testing; Other: Olfaction testing; Diagnostic Test: Spirometry; Other: Walk Test

INTERVENTIONS:
Diagnostic Test: MRI (heart, brain, lungs, liver) — MRI (heart, brain, lungs, liver)
Diagnostic Test: Bloodwork — Serum biomarkers to assess systemic inflammation, renal function, cardiac injury, liver injury and steatosis, ACE-2 related peptides, cytokines, Activin A and autoantibodies to cardiac antigens, humoral cell RNA
Other: Cognitive testing — NIH toolbox Cognitive Measures
Other: Olfaction testing — Brief Smell Identification Test (BSIT)
Diagnostic Test: Spirometry — Spirometry to evaluate forced expiratory volume in 1 second and forced vital capacity
Other: Walk Test — Walk test to record overall distance walked in 6 minutes and time taken to walk the first 25 feet

SUMMARY:
While many people with COVID-19 suffer from respiratory disease, there is growing evidence that the virus also affects other organs. The purpose of this study is to better understand the effects of COVID-19 on the lungs and other organs.

The study investigators have developed new techniques in Magnetic Resonance Imaging (MRI) to scan the lungs, heart, brain and liver. The study investigators hope to learn more about how the virus causes inflammation in these organs and how this inflammation changes over time as people recover from COVID-19 illness.

The study aims to enroll 228 people in Alberta. Participants will undergo one or more MRI scans and have blood testing at one or more time points to assess for inflammation, kidney function, liver function and possible heart injury. Participants will also undergo testing to assess sense of smell, cognition (thinking and memory), spirometry (breathing test for lung function) and and exercise tolerance (walk test).

The study investigators hope this study will help us learn more about the long-term risks of COVID-19 disease.

DETAILED DESCRIPTION:
Participants with newly or recently diagnosed COVID-19 infection (inpatients and outpatients) will undergo multi-organ MRI (heart, brain, lungs, liver), blood work, and functional testing at one or more time points. Functional testing will include olfaction testing, cognitive testing, spiromety, and a walk test.

ELIGIBILITY:
Troponin substudy Inclusion Criteria:

1. 18 years of age or older
2. Willing and able to provide informed consent
3. COVID-19 positive test (within 14 days of positive test date)
4. High-sensitivity Troponin-I >100ng/L or Troponin T > 52ng/L
5. Ability to obtain Baseline MRI imaging within 7 days (up to 14 days maximum) of Troponin result

Troponin substudy Exclusion Criteria:

1. Contraindication to MRI or MRI contrast
2. GFR < 30ml/kg/min/1.73m2
3. Hemodynamic instability requiring inotropic agents
4. Active ventilatory support

Late cross-sectional substudy Inclusion Criteria:

1. 18 years of age or older
2. Willing and able to provide informed consent
3. Previously diagnosed with COVID-19 > 3 months ago
4. Ability to obtain MRI imaging at minimum 12 weeks from COVID-19 diagnosis

Late cross-sectional substudy Exclusion Criteria:

1. Contraindication to MRI or MRI contrast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with new or recent COVID-19 infection.
Sampling Method: Non-Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2021-09-22 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Native myocardial T1 relaxation time | 12 weeks post COVID-19 diagnosis
  Myocardial T1 is a surrogate marker of myocardial edema and the most sensitive MRI measure of acute myocarditis. We will show that myocardial T1 at baseline is significantly higher than myocardial T1 at 12 weeks follow-up. At 12 weeks, we will also compare native myocardial T1 in patients with baseline elevated troponin to those with baseline normal troponin as well as healthy controls

SECONDARY OUTCOMES:
FLAIR imaging | 12 weeks post COVID-19 diagnosis
  Similar within group and between group comparisons of MRI derived lung water content, liver water content, and the presence of brain inflammation on FLAIR imaging
Compare 12-week cognitive testing to the corresponding findings on MRI of brain, heart and lung at baseline | 12 weeks post COVID-19 diagnosis
  Compare 12-week cognitive testing (NIH toolbox score) to the corresponding findings on MRI of brain, heart and lung at baseline
Compare 12-week spirometry to the corresponding findings on MRI of brain, heart and lung at baseline | 12 weeks post COVID-19 diagnosis
  Compare 12-week spirometry (FEV1, FVC and FEV1:FVC) to the corresponding findings on MRI of brain, heart and lung at baseline
Compare 12-week walk test results to the corresponding findings on MRI of brain, heart and lung at baseline | 12 weeks post COVID-19 diagnosis
  Compare 12-week walk test results (distance and time) to the corresponding findings on MRI of brain, heart and lung at baseline
Compare 12-week cognitive testing in patients with normal smell and/or normal appearing brainstem on MRI to patients with no or impaired smell and/or injury to brainstem on MRI | 12 weeks post COVID-19 diagnosis
  Compare 12-week cognitive testing in patients with normal smell and/or normal appearing brainstem on MRI to patients with no or impaired smell and/or injury to brainstem on MRI
Compare MRI measures of organ dysfunction at 12-24 weeks in survivors according to severity of prior COVID-19 illness: (i) hospitalized, (ii) symptomatic, not hospitalized and (iii) asymptomatic | 12-24 weeks post COVID-19 diagnosis
  Compare MRI measures of organ dysfunction at 12-24 weeks in survivors according to severity of prior COVID-19 illness: (i) hospitalized, (ii) symptomatic, not hospitalized and (iii) asymptomatic

CONTACTS AND LOCATIONS:
Overall Officials: Ian Paterson, MD, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Paterson DI, White JA, Beaulieu C, Sherrington R, Prado CM, Tandon P, Halloran K, Smith S, McCombe JA, Ritchie B, Pituskin E, Haykowsky MJ, Coulden R, Emery D, Tsui AK, Wu KY, Oudit GY, Ezekowitz JA, Thompson RB. Rationale and design of the multi organ inflammation with serial testing study: a comprehensive assessment of functional and structural abnormalities in patients with recovered COVID-19. Front Med (Lausanne). 2024 Jul 24;11:1392169. doi: 10.3389/fmed.2024.1392169. eCollection 2024. PMID 39114821
- [Derived] Crosier R, Kafil TS, Paterson DI. Imaging for Cardiovascular Complications of COVID-19: Cardiac Manifestations in Context. Can J Cardiol. 2023 Jun;39(6):779-792. doi: 10.1016/j.cjca.2023.01.022. Epub 2023 Jan 31. PMID 36731604